CLINICAL TRIAL: NCT05624580
Title: Investigation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Injections of NNC0582-0001 in Healthy Adults
Brief Title: A Study to Look at Safety and Tolerability of NNC0582-0001, How it is Transported Throughout the Body and How it Works in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6582-4838; U1111-1274-4316 (Other: World Health Organization (WHO)); 2022-001813-38 (EudraCT Number); 2023-506928-83 (Registry Identifier: European Medical Agency (EMA))
Record Dates: First submitted 2022-11-08; First posted 2022-11-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single Dose 1: NNC0582-0001 10 milligram (mg) (Experimental): Participants will receive a single dose of NNC0582-0001 10 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0582-0001; Drug: Placebo
- Single Dose 2: NNC0582-0001 30 mg (Experimental): Participants will receive a single dose of NNC0582-0001 30 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0582-0001; Drug: Placebo
- Single Dose 3: NNC0582-0001 90 mg (Experimental): Participants will receive a single dose of NNC0582-0001 90 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0582-0001; Drug: Placebo
- Single Dose 4: NNC0582-0001 250 mg (Experimental): Participants will receive a single dose of NNC0582-0001 250 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0582-0001; Drug: Placebo
- Single Dose 5: NNC0582-0001 600 mg (Experimental): Participants will receive a single dose of NNC0582-0001 600 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0582-0001; Drug: Placebo
- Single Dose 6: NNC0582-0001 1000 mg (Experimental): Participants will receive a single dose of NNC0582-0001 1000 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0582-0001; Drug: Placebo

INTERVENTIONS:
Drug: NNC0582-0001 — Participants will receive single dose of any of the six dose levels of subcutaneous NNC0582-0001 in a sequential manner with the dose increasing between cohorts.
Drug: Placebo — Participants will receive single dose of subcutaneous injection of placebo matched to NNC0582-0001.

SUMMARY:
This is a single-center, randomized, double-blind, sequential-group, placebo-controlled study with six sequential single dose cohorts with ascending dose levels in healthy adult participants. This study will assess the safety, tolerability, the pharmacokinetics from single subcutaneous administrations of NNC0582-0001 and explores the pharmacodynamics in healthy participants. Participants will be randomized in a 3:1 ratio to receive a fixed single dose (1-day) of NNC0582 0001 or placebo by injections under the skin. Participants will be followed up for 52 weeks post dose.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential or male aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) from 20.0 to 30.0 kilogram per square meter (kg/m^2) (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram, and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Glycated haemoglobin (HbA1c) greater than or equal to 5.7 percent (39 millimoles per mole [mmol/mol]) at screening.
* Any of the below laboratory safety parameters at screening outside normal range, see laboratory provided reference ranges for specific values (re-screening or re-sampling is NOT allowed if the participant has failed one of the exclusion criteria related to laboratory parameters):
* Alanine aminotransferase (ALT)
* Aspartate aminotransferase (AST)
* Bilirubin
* Estimated glomerular filtration rate (eGFR) below 90 milliliters per minute per 1.73m^2 (mL/min/1.73m^2)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From dosing (Day 1) until End of Study visit (Week 52)
  Measured as number of events.

SECONDARY OUTCOMES:
AUC0-∞: The area under the NNC0582-0001 plasma concentration-time curve from time zero to infinity after a single dose. | From dosing (Day 1) to 168 hours after dosing
  Measured in hours * nanogram per mililiter (h*ng/mL).
Cmax: The maximum concentration of NNC0582-0001 in plasma | From dosing (Day 1) to 168 hours after dosing
  Measured in nanogram per mililiter (ng/mL).
tmax: The time from dose administration to maximum plasma concentration of NNC0582-0001 | From dosing (Day 1) to 168 hours after dosing
  Measured in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Clinical Trials Unit / Center for Medical Research, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.